CLINICAL TRIAL: NCT04621474
Title: The Utility of Non-magnified NBI in Barrett's Oesophagus Neoplasia Detection and Delineation by Non-expert Endoscopists
Brief Title: Non-magnified NBI in Barrett's Oesophagus Neoplasia Detection and Delineation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Massimiliano di Pietro, MD, Senior Clinician Scientist, University of Cambridge
Other Study IDs: NiBOD
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Narrow Band Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Narrow band imaging (NBI) — Narrow-band imaging uses specific light wavelengths of 415 nm (blue) and 540 nm (green) due to a special filter which is electronically activated by a switch in the endoscope.
  Other Names: Non-magnified white-light endoscopy (WLE)

SUMMARY:
Endoscopy plays a pivotal role in the management (diagnosis and treatment) of Barrett's related neoplasia. The standard endoscopy is generally done under white light, which is known to be imperfect in detecting early neoplastic lesion. Narrow band imaging (NBI) improves definition of the superficial morphology and vasculature of GI mucosa. Some studies have shown the potential to improve diagnostic accuracy and reduce the number of biopsies required for Barrett's related neoplasia. This can ultimately improve the cost-effectiveness of endoscopic surveillance. The ability to discriminate between healthy and diseased tissue also makes NBI a useful technique for the delineation of lesions to treat with endoscopic mucosal resection (EMR). However not all studies provide evidence of diagnostic utility. Also the majority of these studies have been conducted by expert endoscopists, which makes the results difficult to extend to general endoscopy practice. The limited number of Barrett's specialists in certain areas of the country validates the need for a study to investigate whether there is an objective improvement in detection and delineation of Barrett's neoplastic lesions by less experienced observers. The aim of this study was to determine the utility of non-magnified NBI in non-expert identification of lesions as compared to expert endoscopists as well as the inter-observer agreement among endoscopists on WLE and NBI.

DETAILED DESCRIPTION:
Matched non-magnified white-light endoscopy (WLE) and narrow band imaging (NBI) images of Barrett's oesophagus with and without lesions from the same level will be obtained prospectively. Lesions will be delineated by 3 expert endoscopists and the overlap between all delineations for each image, regarded as the "sweet spot", will be used as the gold standard. The images will then be assessed by a group of non-expert endoscopists (trainees and nurse endoscopists) as well as senior endoscopists with no interest in Barrett's. First, white light images will be assessed, followed by a wash-out period and then NBI. Assessments will be carried out using a computer application designed in MATLAB. Observers will be also asked to complete the following 1) Paris classification of lesion 2) delineation of the lesion on the screen 3) rate the ability to delineate the lesion for each of the two respective imaging modalities (using a Visual analog scale (VAS score 1-10), 4) choice a single point for virtual diagnostic biopsy. Thus, the quantitative interobserver agreement of the delineations for WLE and NBI will be calculated. VAS scores for the ability to delineate the lesion will be compared between WLE and NBI. Rate of inclusion of the biopsy point in the sweet spot on WLE and NBI will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with dysplastic or non-dysplastic BO at least C1 or M2 in length

Exclusion Criteria:

* Reflux oesophagitis (Los Angeles grade ≥C);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surveillance for Barrett's oesophagus or work up for Barrett's related neoplasia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-04-08 (Estimated); Study Completion 2021-04-08 (Estimated)

PRIMARY OUTCOMES:
Lesion identification | 1 year
  Identification of lesions by non Barrett's expert endoscopists on WLE and non-magnified NBI as compared to expert endoscopists
Inter-observer agreement | 1 year
  Inter-observer agreement among endoscopists on WLE and NBI

SECONDARY OUTCOMES:
Preferred imaging modality | 1 year
  Preferred imaging modality for assessment of Barrett's by endoscopists

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano di Pietro, MD, Principal Investigator — MRC Cancer Unit.University of Cambridge.
Locations (1):
- MRC Cancer Unit, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sami SS, Subramanian V, Butt WM, Bejkar G, Coleman J, Mannath J, Ragunath K. High definition versus standard definition white light endoscopy for detecting dysplasia in patients with Barrett's esophagus. Dis Esophagus. 2015 Nov-Dec;28(8):742-9. doi: 10.1111/dote.12283. Epub 2014 Sep 10. PMID 25209721
- [Background] Swager AF, Curvers WL, Bergman JJ. Diagnosis by Endoscopy and Advanced Imaging of Barrett's Neoplasia. Adv Exp Med Biol. 2016;908:81-98. doi: 10.1007/978-3-319-41388-4_5. PMID 27573768
- [Result] Sharma P, Hawes RH, Bansal A, Gupta N, Curvers W, Rastogi A, Singh M, Hall M, Mathur SC, Wani SB, Hoffman B, Gaddam S, Fockens P, Bergman JJ. Standard endoscopy with random biopsies versus narrow band imaging targeted biopsies in Barrett's oesophagus: a prospective, international, randomised controlled trial. Gut. 2013 Jan;62(1):15-21. doi: 10.1136/gutjnl-2011-300962. Epub 2012 Feb 7. PMID 22315471
- [Result] Yoshida T, Inoue H, Usui S, Satodate H, Fukami N, Kudo SE. Narrow-band imaging system with magnifying endoscopy for superficial esophageal lesions. Gastrointest Endosc. 2004 Feb;59(2):288-95. doi: 10.1016/s0016-5107(03)02532-x. PMID 14745410
- [Result] de Groof AJ, Swager AF, Pouw RE, Weusten BLAM, Schoon EJ, Bisschops R, Pech O, Meining A, Neuhaus H, Curvers WL, Bergman JJGHM. Blue-light imaging has an additional value to white-light endoscopy in visualization of early Barrett's neoplasia: an international multicenter cohort study. Gastrointest Endosc. 2019 Apr;89(4):749-758. doi: 10.1016/j.gie.2018.10.046. Epub 2018 Nov 9. PMID 30419218